CLINICAL TRIAL: NCT05935124
Title: A Randomized Comparison Between White Light Endoscopy (WLE) and Bright Narrow Band Imaging (B-NBI) in the Diagnosis of Right Sided Colonic Polyps in Asymptomatic Subjects Undergoing Screening Colonoscopy
Brief Title: White Light vs Narrow Band Imagingin the Diagnosis of Right Sided Colonic Polyps in Asymptomatic Subjects Undergoing Screening Colonoscopy
Acronym: WLEvsB-NBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Endoscopy, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4222
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Adenoma Colon

STUDY DESIGN:
Intervention Model Description: randomized crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First withdrawal - White light endoscopy (Other): white light (WLE) high definition colonoscope (Olympus 190 series) first and then B-NBI
  Interventions: Diagnostic Test: WLE first, then B-NBI
- First withdrawal - Bright Narrow Band Imagin (Other): B-NBI first and then WLE with the same colonoscope.
  Interventions: Diagnostic Test: WLE first, then B-NBI

INTERVENTIONS:
Diagnostic Test: WLE first, then B-NBI

SUMMARY:
A randomized controlled crossover study to determine if narrow band imaging or white light endoscopy is superior in detecting right colonic polyps in average risk subjects undergoing screening colonoscopy

DETAILED DESCRIPTION:
Removal of colorectal adenomas prevents occurrence of cancers. It is recognized that colonoscopy can miss colorectal adenomas and early cancers. Proximal colon polyp detection rate is lower compared to distal colon detection rates. This may be partially due to the higher prevalence of flat polyps and sessile serrated adenomas (SSAs) which are harder to visualize. There is a need to further improve performance of colonoscopy. A second evaluation of the right colon within the same procedure may yield an additional detection rate of 5-10%, however retro-flexion has not proven to be superior to a second forward viewing examination. The use of chromo-endoscopy has been shown to improve detection of flat adenomas. Narrow band imaging was introduced in year 2006. It is similar to chromo-endoscopy in that it provides more mucosal details. This enables endoscopists to accurately describe the pit pattern of adenomas. NBI has been used as a substitute to chromo-endoscopy. In pooled analysis, NBI is comparable to chromo-endoscopy in their sensitivity and specificity in the diagnosis of malignant colorectal adenomas. Unfortunately, the use of NBI has not been shown to conclusively improve rate of colorectal adenoma detection. Two of 3 randomized trials that compared WLE to NBI showed a higher adenoma detection rate with the use of NBI. In a study by Rex et al., the rate was however similar with either modality. In a pooled analysis, NBI was only marginally better than WLE.

The effective use of NBI depends on the quality of bowel preparation and the experience of endoscopist. In the presence of fecal matters, NBI tends to be dark and detection of small adenomas becomes difficult. The prototype bright NBI coupled with high definition resolution is likely to overcome this drawback of original NBI.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects undergoing screening colonoscopy
* age > 50.
* average risk subjects defined as those without a personal history of inflammatory bowel disease, colon adenoma or cancer or family history of FAP or Familial non-polyposis syndrome or first degree relatives having diagnosed to have colo-rectal carcinoma, no colonoscopy in past 5 years and, ability to provide a written consent to trial participation

Exclusion Criteria:

* unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rate of right sided polyp detection with WLE and B-NBI | 1 day

SECONDARY OUTCOMES:
Rate of the detection of SSPs in the right colon with WLE and B-NBI | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No